CLINICAL TRIAL: NCT00726323
Title: A Phase II Study of the c-MET RTK Inhibitor XL880 in Subjects With Papillary Renal-Cell Carcinoma
Brief Title: A Phase II Study of GSK1363089 (Formerly XL880) for Papillary Renal-Cell Carcinoma (PRC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MET111644; NCT00345423 (obsolete NCT alias)
Record Dates: First submitted 2008-07-29; First posted 2008-07-31 (Estimated); Results first posted 2017-12-11 (Actual); Last update posted 2017-12-11 (Actual); Status verified 2017-09

CONDITIONS: Carcinoma, Renal Cell
Keywords: c-Met; Papillary Renal Cell Carcinoma(PRC); Sporadic papillary renal cell carcinoma,; Clear cell renal carcinoma; Hereditary papillary renal cell carcinoma,
MeSH Terms: conditions — Carcinoma, Renal Cell; Papillary renal cell carcinoma, sporadic | interventions — GSK 1363089

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 5/9 dosing (Experimental): 240 mg of foretinib on a 5 day on / 9 day off regimen every 14 days.
  Interventions: Drug: foretinib (formerly GSK1363089 or XL880)
- daily dosing (Experimental): 80 mg foretinib on a daily dosing regimen
  Interventions: Drug: foretinib (formerly GSK1363089 or XL880)

INTERVENTIONS:
Drug: foretinib (formerly GSK1363089 or XL880) — treatment with oral foretinib on one of 2 dosing regimens: 240 mg on a 5 day on / 9 day off schedule every 14 days, or 80 mg on a daily dosing schedule
  Other Names: GSK1363089 (formerly XL880)

SUMMARY:
This clinical study is being conducted at multiple sites to determine the best confirmed response rate, safety, and tolerability of GSK1363089 treatment in papillary renal cell carcinoma. Papillary renal cell carcinoma may be classified into hereditary and sporadic forms; subjects with either classification will be accepted into this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of PRC with metastatic disease or bilateral multifocal renal tumors localized to kidneys. Measurable disease, ECOG performance status of </= 2.
* Adequate bone marrow reserve, hepatic, renal, and cardiovascular function.

Exclusion Criteria:

* Radiation to >/=25% of bone marrow within 14 days of GSK1363089, more than 1 prior anti-cancer therapy, received prior treatment with a c-met inhibitor, brain metastases,
* Any uncontrolled intercurrent illness,
* Pregnant or breastfeeding,
* HIV positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2006-06-30 (Actual); Primary Completion 2010-08-18 (Actual); Study Completion 2010-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (12):
- United States (12):
  - GSK Investigational Site, Greenbrae, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Stanford, California
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Bethesda, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, New Brunswick, New Jersey
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Choueiri TK, Vaishampayan U, Rosenberg JE, Logan TF, Harzstark AL, Bukowski RM, Rini BI, Srinivas S, Stein MN, Adams LM, Ottesen LH, Laubscher KH, Sherman L, McDermott DF, Haas NB, Flaherty KT, Ross R, Eisenberg P, Meltzer PS, Merino MJ, Bottaro DP, Linehan WM, Srinivasan R. Phase II and biomarker study of the dual MET/VEGFR2 inhibitor foretinib in patients with papillary renal cell carcinoma. J Clin Oncol. 2013 Jan 10;31(2):181-6. doi: 10.1200/JCO.2012.43.3383. Epub 2012 Dec 3. PMID 23213094
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: MET111644 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: MET111644 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: MET111644 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: MET111644 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: MET111644 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: MET111644 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted from 30 June 2006 till 18 August 2010 across 10 centers in the United States (US). A total of 60 participants with papillary renal-cell carcinoma (PRC) were planned to be enrolled.
Pre-assignment Details: A total of 74 participants with PRC were enrolled in the study.
Groups:
- Intermittent 5 & 9 Dosing Regimen: Eligible participants received oral foretinib bisphosphate 240 milligrams (mg) on Days 1 to 5 of every 14-day cycle. Participants continued this schedule for 8 weeks. The treatment drug was supposed to be stopped any time in case of disease progression. All participants were followed-up up to 8 weeks after the last dose of the study drug for tumor assessment.
- Daily Dosing Regimen: Eligible participants received oral foretinib bisphosphate 80 mg daily of every 14-day cycle. Participants continued this schedule for 8 weeks. treatment drug was supposed to be stopped any time in case of disease progression. All participants were followed-up up to 8 weeks after the last dose of the study drug for tumor assessment.
Period: Overall Study
Arm/Group | Intermittent 5 & 9 Dosing Regimen | Daily Dosing Regimen
Started | 37 | 37
Completed | 0 | 6
Not Completed | 37 | 31
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Progressive disease | 23 | 16
Not completed — Clinical progression | 0 | 3
Not completed — Adverse Event | 9 | 9
Not completed — Death | 1 | 0
Not completed — Participant wished to discontinue | 0 | 1
Not completed — Metastatic lesions inferred cyst | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Safety population included all participants who passed the screening criteria, were enrolled in the study and received at least one dose of the study drug.
Groups:
- Intermittent 5 & 9 Dosing Regimen: Eligible participants received oral foretinib bisphosphate 240 mg on Days 1 to 5 of every 14-day cycle. Participants continued this schedule for 8 weeks. The treatment drug was supposed to be stopped any time in case of disease progression. All participants were followed-up up to 8 weeks after the last dose of the study drug for tumor assessment.
- Total: Total of all reporting groups
Arm/Group | Intermittent 5 & 9 Dosing Regimen | Daily Dosing Regimen | Total
Number analyzed (Participants) | 37 | 37 | 74
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.1 (11.84) | 56.2 (14.32) | 55.6 (13.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 30 | 29 | 59
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 1 | 2
  Black or African American | 2 | 3 | 5
  White | 32 | 32 | 64
  Multiple | 0 | 1 | 1
  Other | 1 | 0 | 1
  Unknown | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors (RECIST) Criteria Version 1.0
Description: Overall response rate is the percentage of participants for whom the best overall response to the study drug was a confirmed partial response (PR) or confirmed complete response (CR). Best overall response and its associated confirmation criteria, RECIST; Version 1.0) was based on the Investigator's assessment of the target and non target lesions.
Time Frame: At the end of forth year
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Intermittent 5 & 9 Dosing Regimen | Daily Dosing Regimen
Number analyzed (Participants) | 37 | 37
Percentage of participants | 13.5 [4.5 to 28.8] | 13.5 [4.5 to 28.8]

2. Secondary Outcome: Disease Stabilization Rate Over Period
Description: The percentage of participants for whom the best overall response was a confirmed PR, confirmed CR, or stable disease. Exact confidence intervals were obtained using the Clopper-Pearson method. Exact confidence intervals were obtained using the Clopper-Pearson method.
Time Frame: Up to 4 years
Population: Safety population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Intermittent 5 & 9 Dosing Regimen | Daily Dosing Regimen
Number analyzed (Participants) | 37 | 37
Percentage of participants | 91.9 [78.1 to 98.3] | 83.8 [68.0 to 93.8]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression free survival is defined as the time between the date of first dose of study drug and the date of the first occurrence of either tumor progression per RECIST or clinical assessment of progression as assessed by Investigator or Death due to any cause, whichever occurs the first. For participants who did not reach an event (disease progression or death) at the time of data cutoff, PFS was censored at the date of the last available tumor measurement. For participants who did not have any post-baseline tumor assessments, PFS was right censored at Day 1. For any participants who received subsequent anticancer therapy, PFS was right censored at the date of last adequate tumor assessment on or prior to the date of anticancer initiation. For any participants, who died or progressed after an extended follow-up, PFS was censored at the date of last adequate assessment prior to the extended loss to follow-up.
Time Frame: At the end of forth year
Population: Safety population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Intermittent 5 & 9 Dosing Regimen | Daily Dosing Regimen
Number analyzed (Participants) | 37 | 37
Months | 11.56 [5.78 to 16.99] | 9.07 [5.78 to 10.91]

4. Secondary Outcome: Time to Response (TTR) Over Period
Description: Time to response is the time between the date of first dose of study drug and the date of first response (for participants who had overall responses that were later confirmed as CR/PR). For the 6 participants in the daily dosing cohort who did not reach a response as of data cutoff, the time to response was censored at the date of the last visit. The median time to response was not estimable in either of the dosing cohorts or in the overall safety population using the Kaplan-Meier method.
Time Frame: Up to 4 years
Population: Safety population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Intermittent 5 & 9 Dosing Regimen | Daily Dosing Regimen
Number analyzed (Participants) | 37 | 37
Months | NA [22.05 to NA] — The median time to response was not estimable. | NA [12.88 to NA] — The median time to response was not estimable.

5. Secondary Outcome: Duration of Response (DOR)
Description: Duration of response is defined as the time between the date of first response (later confirmed CR or confirmed PR) and the date of the first occurrence of one of the events as tumor progression per RECIST as assessed by Investigator, termination of the study drug due to disease progression, death due to any cause, disease progression as documented on the follow-up or participant status form Initiation of subsequent anticancer therapy. For the 6 participants in the daily dosing cohort who did not reach a response as of data cutoff, the duration of response was censored at the date of the last available tumor measurement.
Time Frame: Up to 4 years
Population: Safety Population- All Objective Responders (those who did not reach an event by the time of data cut-off as defined in protocol)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Intermittent 5 & 9 Dosing Regimen | Daily Dosing Regimen
Number analyzed (Participants) | 5 | 5
Months | 20.50 [5.55 to 20.50] | 18.46 [5.55 to 18.46]

6. Secondary Outcome: Duration of Stable Disease (SD)
Description: Duration of SD is defined as the time between the date of first dose of study drug and the date of the first occurrence of one of the tumor progression per RECIST as assessed by Investigator, termination of the study drug due to disease progression, death due to disease progression, or disease progression as documented on the follow-up participants status form Initiation of subsequent anticancer therapy. For the 6 participants in the daily dosing cohort who did not reach a response as of data cutoff, the duration of stable disease was right censored at the date of the last available tumor measurement.
Time Frame: Up to 4 years
Population: Safety population. All participants with Best overall response, not progressive disease were considered.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Intermittent 5 & 9 Dosing Regimen | Daily Dosing Regimen
Number analyzed (Participants) | 34 | 31
Months | 12.88 [6.14 to 16.99] | 9.26 [7.16 to 10.84]

7. Secondary Outcome: Overall Survival
Description: Overall survival, which is defined as the time between the date of first dose of study drug and the date of death (due to any cause). For participants who were alive at the time of data cutoff, duration of overall survival was right censored at the date of last contact. Duration of overall survival = date of death/censoring - date of first dose +1. Percentiles and confidence intervals are calculated using Kaplan-Meier methods.
Time Frame: Up to 4 years
Population: Safety population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Intermittent 5 & 9 Dosing Regimen | Daily Dosing Regimen
Number analyzed (Participants) | 37 | 37
Months | NA [11.83 to NA] — The median survival time was not estimable. | NA [NA to NA] — The median survival time was not estimable.

8. Secondary Outcome: Number of Participants With Change in Common Terminology Criteria for Adverse Events (CTCAE) Grade of Clinical Chemistry Parameters Over Period
Description: The worst case overall common terminology criteria for adverse events (CTCAE) grade shift post Baseline for each parameter was mentioned. Only worst case scenarios are presented. CTCAE grading was done as per intensity namely mild moderate severe life-threatening or Death. Analysis was done for Alanine aminotransferases (ALT), aspartate aminotransferases (AST), Albumin, alkaline phosphatase (ALP), calcium, sodium, potassium, glucose, amylase, carbon dioxide, phosphate, gamma glutamyl transferases (GGT), and triglycerol lipase. High (H) levels and low (L) levels were measured.
Time Frame: Up to 4 years
Population: Safety population
Measure: Number; unit: Participants
Arm/Group | Intermittent 5 & 9 Dosing Regimen | Daily Dosing Regimen
Number analyzed (Participants) | 37 | 37
Participants
  ALT, Grade 0 to 1: number analyzed (Participants) | 36 | 37
  ALT, Grade 0 to 1 | 24 | 21
  ALT, Grade 0 to 2: number analyzed (Participants) | 36 | 37
  ALT, Grade 0 to 2 | 4 | 1
  ALT, Grade 0 to 3: number analyzed (Participants) | 36 | 37
  ALT, Grade 0 to 3 | 0 | 1
  ALT, Grade 1 to 2: number analyzed (Participants) | 36 | 37
  ALT, Grade 1 to 2 | 1 | 2
  Albumin, Grade 0 to 1: number analyzed (Participants) | 36 | 37
  Albumin, Grade 0 to 1 | 9 | 12
  Albumin, Grade 0 to 2: number analyzed (Participants) | 36 | 37
  Albumin, Grade 0 to 2 | 8 | 11
  Albumin, Grade 0 to 3: number analyzed (Participants) | 36 | 37
  Albumin, Grade 0 to 3 | 1 | 2
  Albumin, Grade 1 to 2: number analyzed (Participants) | 36 | 37
  Albumin, Grade 1 to 2 | 6 | 5
  Albumin, Grade 1 to 3: number analyzed (Participants) | 36 | 37
  Albumin, Grade 1 to 3 | 0 | 1
  ALP, Grade 0 to 1: number analyzed (Participants) | 36 | 37
  ALP, Grade 0 to 1 | 12 | 16
  ALP, Grade 0 to 2: number analyzed (Participants) | 36 | 37
  ALP, Grade 0 to 2 | 1 | 0
  ALP, Grade 0 to 3: number analyzed (Participants) | 36 | 37
  ALP, Grade 0 to 3 | 0 | 0
  ALP, Grade 0 to 4: number analyzed (Participants) | 36 | 37
  ALP, Grade 0 to 4 | 0 | 0
  ALP, Grade 1 to 2: number analyzed (Participants) | 36 | 37
  ALP, Grade 1 to 2 | 0 | 2
  Amylase, Grade 0 to 1: number analyzed (Participants) | 35 | 37
  Amylase, Grade 0 to 1 | 9 | 6
  Amylase, Grade 0 to 2: number analyzed (Participants) | 35 | 37
  Amylase, Grade 0 to 2 | 1 | 2
  Amylase, Grade 0 to 3: number analyzed (Participants) | 35 | 37
  Amylase, Grade 0 to 3 | 1 | 1
  Amylase, Grade 1 to 2: number analyzed (Participants) | 35 | 37
  Amylase, Grade 1 to 2 | 0 | 1
  Amylase, Grade 2 to 3 | 1 | 0
  AST, Grade 0 to 1: number analyzed (Participants) | 36 | 37
  AST, Grade 0 to 1 | 23 | 27
  AST, Grade 0 to 2: number analyzed (Participants) | 36 | 37
  AST, Grade 0 to 2 | 8 | 3
  AST, Grade 0 to 3: number analyzed (Participants) | 36 | 37
  AST, Grade 0 to 3 | 0 | 1
  AST, Grade 1 to 2: number analyzed (Participants) | 36 | 37
  AST, Grade 1 to 2 | 2 | 0
  AST, Grade 2 to 3: number analyzed (Participants) | 36 | 37
  AST, Grade 2 to 3 | 1 | 0
  Blilirubin, Grade 0 to 1: number analyzed (Participants) | 36 | 37
  Blilirubin, Grade 0 to 1 | 7 | 1
  Blilirubin, Grade 0 to 3: number analyzed (Participants) | 36 | 37
  Blilirubin, Grade 0 to 3 | 1 | 0
  Blilirubin, Grade 1 to 2: number analyzed (Participants) | 36 | 37
  Blilirubin, Grade 1 to 2 | 1 | 0
  Carbon di oxide, Grade 0 to 1: number analyzed (Participants) | 36 | 37
  Carbon di oxide, Grade 0 to 1 | 11 | 9
  Creatinine, Grade 0 to 1: number analyzed (Participants) | 36 | 37
  Creatinine, Grade 0 to 1 | 6 | 11
  Creatinine, Grade 0 to 2: number analyzed (Participants) | 36 | 37
  Creatinine, Grade 0 to 2 | 3 | 0
  Creatinine, Grade 0 to 3: number analyzed (Participants) | 36 | 37
  Creatinine, Grade 0 to 3 | 2 | 0
  Creatinine, Grade 1 to 0: number analyzed (Participants) | 36 | 37
  Creatinine, Grade 1 to 0 | 1 | 0
  Creatinine, Grade 1 to 2: number analyzed (Participants) | 36 | 37
  Creatinine, Grade 1 to 2 | 2 | 8
  GGT, Grade 0 to 1: number analyzed (Participants) | 36 | 37
  GGT, Grade 0 to 1 | 7 | 6
  GGT, Grade 1 to 0: number analyzed (Participants) | 36 | 37
  GGT, Grade 1 to 0 | 0 | 0
  GGT, Grade 2 to 0: number analyzed (Participants) | 36 | 0
  GGT, Grade 2 to 0 | 0 |
  GGT, Grade 2 to 1: number analyzed (Participants) | 36 | 0
  GGT, Grade 2 to 1 | 0 |
  Phosphate, Grade 0 to 1: number analyzed (Participants) | 36 | 37
  Phosphate, Grade 0 to 1 | 1 | 1
  Phosphate, Grade 0 to 2: number analyzed (Participants) | 36 | 37
  Phosphate, Grade 0 to 2 | 8 | 10
  Phosphate, Grade 0 to 3: number analyzed (Participants) | 36 | 37
  Phosphate, Grade 0 to 3 | 13 | 8
  Phosphate, Grade 2 to 0: number analyzed (Participants) | 36 | 37
  Phosphate, Grade 2 to 0 | 0 | 1
  Phosphate, Grade 2 to 3: number analyzed (Participants) | 36 | 37
  Phosphate, Grade 2 to 3 | 0 | 1
  Phosphate, Grade 2 to 4 | 1 | 0
  Triglycerol lipase, Grade 0 to 1: number analyzed (Participants) | 36 | 37
  Triglycerol lipase, Grade 0 to 1 | 6 | 9
  Triglycerol lipase, Grade 0 to 2: number analyzed (Participants) | 36 | 37
  Triglycerol lipase, Grade 0 to 2 | 1 | 6
  Triglycerol lipase, Grade 0 to 3: number analyzed (Participants) | 36 | 37
  Triglycerol lipase, Grade 0 to 3 | 4 | 4
  Triglycerol lipase, Grade 0 to 4: number analyzed (Participants) | 36 | 37
  Triglycerol lipase, Grade 0 to 4 | 0 | 1
  Triglycerol lipase, Grade 1 to 3: number analyzed (Participants) | 36 | 37
  Triglycerol lipase, Grade 1 to 3 | 1 | 1
  Triglycerol lipase, Grade 1 to 4: number analyzed (Participants) | 36 | 37
  Triglycerol lipase, Grade 1 to 4 | 1 | 0
  Triglycerol lipase, Grade 2 to 3: number analyzed (Participants) | 37 | 0
  Triglycerol lipase, Grade 2 to 3 | 1 |
  Calcium, L, Grade 0 to 1: number analyzed (Participants) | 36 | 37
  Calcium, L, Grade 0 to 1 | 12 | 14
  Calcium, L, Grade 0 to 2: number analyzed (Participants) | 36 | 37
  Calcium, L, Grade 0 to 2 | 7 | 13
  Calcium, L, Grade 0 to 3: number analyzed (Participants) | 36 | 37
  Calcium, L, Grade 0 to 3 | 1 | 2
  Glucose, L, Grade 0 to 1: number analyzed (Participants) | 36 | 37
  Glucose, L, Grade 0 to 1 | 10 | 11
  Glucose, L, Grade 0 to 2: number analyzed (Participants) | 36 | 37
  Glucose, L, Grade 0 to 2 | 1 | 4
  Glucose, L, Grade 0 to 3: number analyzed (Participants) | 36 | 37
  Glucose, L, Grade 0 to 3 | 0 | 1
  Glucose, L, Grade 1 to 3: number analyzed (Participants) | 36 | 37
  Glucose, L, Grade 1 to 3 | 0 | 1
  Potassium, L, Grade 0 to 1: number analyzed (Participants) | 36 | 37
  Potassium, L, Grade 0 to 1 | 5 | 2
  Potassium, L, Grade 1 to 0: number analyzed (Participants) | 36 | 0
  Potassium, L, Grade 1 to 0 | 1 |
  Sodium, L, Grade 0 to 1: number analyzed (Participants) | 36 | 37
  Sodium, L, Grade 0 to 1 | 11 | 14
  Sodium, L, Grade 0 to 3: number analyzed (Participants) | 36 | 37
  Sodium, L, Grade 0 to 3 | 3 | 6
  Sodium, L, Grade 1 to 3: number analyzed (Participants) | 36 | 0
  Sodium, L, Grade 1 to 3 | 1 |
  Calcium, H, Grade 0 to 1: number analyzed (Participants) | 36 | 37
  Calcium, H, Grade 0 to 1 | 2 | 0
  Glucose, H, Grade 0 to 1: number analyzed (Participants) | 36 | 37
  Glucose, H, Grade 0 to 1 | 16 | 10
  Glucose, H, Grade 0 to 2: number analyzed (Participants) | 36 | 37
  Glucose, H, Grade 0 to 2 | 6 | 4
  Glucose, H, Grade 1 to 0: number analyzed (Participants) | 36 | 37
  Glucose, H, Grade 1 to 0 | 0 | 1
  Glucose, H, Grade 1 to 2: number analyzed (Participants) | 36 | 37
  Glucose, H, Grade 1 to 2 | 4 | 2
  Glucose, H, Grade 1 to 3: number analyzed (Participants) | 36 | 37
  Glucose, H, Grade 1 to 3 | 1 | 0
  Glucose, H, Grade 2 to 3: number analyzed (Participants) | 0 | 37
  Glucose, H, Grade 2 to 3 |  | 1
  Potassium, H, Grade 0 to 1: number analyzed (Participants) | 36 | 37
  Potassium, H, Grade 0 to 1 | 5 | 11
  Potassium, H, Grade 0 to 2: number analyzed (Participants) | 36 | 37
  Potassium, H, Grade 0 to 2 | 8 | 6
  Potaasium, H, Grade 0 to 3: number analyzed (Participants) | 36 | 37
  Potaasium, H, Grade 0 to 3 | 0 | 1
  Potassium, H, Grade 1 to 3: number analyzed (Participants) | 36 | 0
  Potassium, H, Grade 1 to 3 | 1 |
  Sodium, H, Grade 0 to 1: number analyzed (Participants) | 36 | 37
  Sodium, H, Grade 0 to 1 | 6 | 7
  Sodium, H, Grade 1 to 0: number analyzed (Participants) | 0 | 37
  Sodium, H, Grade 1 to 0 |  | 1

9. Secondary Outcome: Number of Participants With Change in CTCAE Grade of Hematological Parameters Over Period (Only Worst Case)
Description: CTCAE gradation The worst case overall CTCAE grade shift post Baseline for each parameter was mentioned. Only worst case scenarios are presented. CTCAE grading was done as per intensity namely mild moderate severe life-threatening or Death. Participants were analyzed for hemoglobin, leukocytes, platelets, percentage of lymphocytes, and percentage of neutrophils.
Time Frame: Up to 4 years
Population: Safety population
Measure: Number; unit: Participants
Arm/Group | Intermittent 5 & 9 Dosing Regimen | Daily Dosing Regimen
Number analyzed (Participants) | 37 | 37
Participants
  Hemoglobin, Grade 0 to 1: number analyzed (Participants) | 36 | 37
  Hemoglobin, Grade 0 to 1 | 12 | 7
  Hemoglobin, Grade 0 to 2: number analyzed (Participants) | 36 | 37
  Hemoglobin, Grade 0 to 2 | 1 | 0
  Hemoglobin, Grade 1 to 2: number analyzed (Participants) | 36 | 37
  Hemoglobin, Grade 1 to 2 | 3 | 2
  Hemoglobin, Grade 1 to 3: number analyzed (Participants) | 36 | 37
  Hemoglobin, Grade 1 to 3 | 1 | 1
  Hemoglobin, Grade 2 to 1: number analyzed (Participants) | 36 | 37
  Hemoglobin, Grade 2 to 1 | 1 | 1
  Leukocytes, Grade 0 to 1: number analyzed (Participants) | 36 | 37
  Leukocytes, Grade 0 to 1 | 5 | 10
  Leukocytes, Grade 0 to 2: number analyzed (Participants) | 36 | 37
  Leukocytes, Grade 0 to 2 | 2 | 0
  Leukocytes, Grade 1 to 2: number analyzed (Participants) | 36 | 0
  Leukocytes, Grade 1 to 2 | 1 |
  Leukocytes, Grade 2 to 0: number analyzed (Participants) | 36 | 0
  Leukocytes, Grade 2 to 0 | 1 |
  Percentage lymphocytes, Grade 0 to 1: number analyzed (Participants) | 36 | 37
  Percentage lymphocytes, Grade 0 to 1 | 5 | 8
  Percentage lymphocytes, Grade 0 to 2: number analyzed (Participants) | 36 | 37
  Percentage lymphocytes, Grade 0 to 2 | 4 | 0
  Percentage lymphocytes, Grade 0 to 3: number analyzed (Participants) | 36 | 37
  Percentage lymphocytes, Grade 0 to 3 | 3 | 2
  Percentage lymphocytes, Grade 1 to 0: number analyzed (Participants) | 36 | 37
  Percentage lymphocytes, Grade 1 to 0 | 0 | 1
  Percentage lymphocytes, Grade 1 to 2: number analyzed (Participants) | 36 | 37
  Percentage lymphocytes, Grade 1 to 2 | 1 | 2
  Percentage lymphocytes, Grade 2 to 0: number analyzed (Participants) | 36 | 37
  Percentage lymphocytes, Grade 2 to 0 | 1 | 0
  Percentage lymphocytes, Grade 2 to 1: number analyzed (Participants) | 36 | 37
  Percentage lymphocytes, Grade 2 to 1 | 0 | 1
  Percentage lymphocytes, Grade 2 to 3: number analyzed (Participants) | 36 | 37
  Percentage lymphocytes, Grade 2 to 3 | 3 | 0
  Percentage lymphocytes, Grade 3 to 4: number analyzed (Participants) | 36 | 0
  Percentage lymphocytes, Grade 3 to 4 | 1 |
  Percentage neutrophils, Grade 0 to 1: number analyzed (Participants) | 36 | 37
  Percentage neutrophils, Grade 0 to 1 | 4 | 4
  Percentage neutrophils, Grade 0 to 2: number analyzed (Participants) | 36 | 37
  Percentage neutrophils, Grade 0 to 2 | 1 | 1
  Percentage neutrophils, Grade 0 to 4: number analyzed (Participants) | 36 | 37
  Percentage neutrophils, Grade 0 to 4 | 0 | 1
  Percentage neutrophils, Grade 1 to 0: number analyzed (Participants) | 36 | 37
  Percentage neutrophils, Grade 1 to 0 | 1 | 0
  Platelets, Grade 0 to 1: number analyzed (Participants) | 36 | 37
  Platelets, Grade 0 to 1 | 12 | 18
  Platelets, Grade 0 to 2: number analyzed (Participants) | 36 | 37
  Platelets, Grade 0 to 2 | 1 | 2
  Platelets, Grade 1 to 2: number analyzed (Participants) | 0 | 37
  Platelets, Grade 1 to 2 |  | 1

10. Secondary Outcome: Number of Participants With Adverse Events, Serious Adverse Events, and Deaths
Description: Adverse event (AE) is an unfavorable change in the health of a participant, including abnormal laboratory findings, that happens during a clinical study or within a certain time period after the study has ended. This change may or may not be caused by the intervention being studied. Serious adverse event (SAE) is an adverse event that results in death, is life-threatening, requires inpatient hospitalization or extends a current hospital stay, results in an ongoing or significant incapacity or interferes substantially with normal life functions, or causes a congenital anomaly or birth defect. Medical events that do not result in death, are not life-threatening, or do not require hospitalization may be considered serious adverse events if they put the participant in danger or require medical or surgical intervention to prevent one of the results listed above.
Time Frame: Up to 4 years
Population: Safety population
Measure: Number; unit: Participants
Arm/Group | Intermittent 5 & 9 Dosing Regimen | Daily Dosing Regimen
Number analyzed (Participants) | 37 | 37
Participants
  Any AE | 37 | 37
  Any SAE | 20 | 22
  Death | 14 | 6

ADVERSE EVENTS:
Time Frame: Approximately up to 48 months
Description: The Safety population included all participants who passed the screening criteria, are enrolled in the study and received at least one dose of the study drug.
Groups:
- Intermittent 5 & 9 Dosing Regimen: Eligible participants received oral foretinib bisphosphate 240 mg on Days 1 to 5 of every 14-day cycle. Participants continued this schedule for 8 weeks. The treatment drug was supposed to be stopped any time in case of disease progression. All participants were followed-up every 8 weeks for tumor assessment, while the participant remained in the treatment extension period.
- Daily Dosing Regimen: Eligible participants received oral foretinib bisphosphate 80 mg daily of every 14-day cycle. Participants continued this schedule for 8 weeks. treatment drug was supposed to be stopped any time in case of disease progression. All participants were followed-up every 8 weeks for tumor assessment, while the participant remained in the treatment extension period.
Arm/Group | Intermittent 5 & 9 Dosing Regimen | Daily Dosing Regimen
All-Cause Mortality (participants affected / at risk) | 14/37 | 6/37
Serious Adverse Events (participants affected / at risk) | 20/37 | 22/37
Other Adverse Events (participants affected / at risk) | 37/37 | 37/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intermittent 5 & 9 Dosing Regimen (N=37) | Daily Dosing Regimen (N=37)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Colour blindness (Congenital, familial and genetic disorders) | 0 | 1
Diplopia (Eye disorders) | 0 | 2
Night blindness (Eye disorders) | 4 | 4
Optic ischaemic neuropathy (Eye disorders) | 0 | 1
Retinal vein occlusion (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 0 | 1
Vitreous haemorrhage (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Disease progression (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 0 | 1
Peridiverticular abscess (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0
Lipase increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebral microhaemorrhage (Nervous system disorders) | 1 | 0
Visual field defect (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 2
Suicidal ideation (Psychiatric disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 2
Renal failure (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Renal haemorrhage (Renal and urinary disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Deep vein thrombosis (Vascular disorders) | 2 | 1
Hypertension (Vascular disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intermittent 5 & 9 Dosing Regimen (N=37) | Daily Dosing Regimen (N=37)
Diarrhoea (Gastrointestinal disorders) | 21 | 29
Nausea (Gastrointestinal disorders) | 28 | 19
Vomiting (Gastrointestinal disorders) | 22 | 13
Constipation (Gastrointestinal disorders) | 14 | 11
Flatulence (Gastrointestinal disorders) | 9 | 5
Abdominal pain (Gastrointestinal disorders) | 6 | 6
Dyspepsia (Gastrointestinal disorders) | 6 | 5
Dry mouth (Gastrointestinal disorders) | 5 | 3
Abdominal distension (Gastrointestinal disorders) | 4 | 3
Abdominal pain upper (Gastrointestinal disorders) | 6 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 5
Abdominal pain lower (Gastrointestinal disorders) | 2 | 2
Ascites (Gastrointestinal disorders) | 1 | 3
Glossodynia (Gastrointestinal disorders) | 2 | 1
Haemorrhoids (Gastrointestinal disorders) | 3 | 0
Stomatiti (Gastrointestinal disorders) | 3 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 2
Fatigue (General disorders) | 31 | 27
Oedema peripheral (General disorders) | 11 | 17
Chills (General disorders) | 7 | 0
Localised oedema (General disorders) | 2 | 2
Pyrexia (General disorders) | 4 | 0
Early satiety (General disorders) | 2 | 1
Pain (General disorders) | 2 | 1
Mucosal inflammation (General disorders) | 2 | 0
Non-cardiac chest pain (General disorders) | 2 | 0
Temperature intolerance (General disorders) | 0 | 2
Hypertension (Vascular disorders) | 28 | 34
Flushing (Vascular disorders) | 2 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 18 | 14
Hypophosphataemia (Metabolism and nutrition disorders) | 11 | 13
Hyperkalaemia (Metabolism and nutrition disorders) | 6 | 5
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 5
Dehydration (Metabolism and nutrition disorders) | 4 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 5
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 2
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 2
Blood creatinine increased (Investigations) | 9 | 6
Aspartate aminotransferase increased (Investigations) | 10 | 4
Lipase increased (Investigations) | 7 | 7
Weight decreased (Investigations) | 6 | 8
Alanine aminotransferase increased (Investigations) | 9 | 4
Blood amylase increased (Investigations) | 5 | 2
Blood lactate dehydrogenase increased (Investigations) | 4 | 3
Electrocardiogram QT prolonged (Investigations) | 0 | 5
Blood urea increased (Investigations) | 3 | 0
Blood alkaline phosphatase increased (Investigations) | 2 | 0
Blood bilirubin increased (Investigations) | 2 | 0
Blood thyroid stimulating hormone increased (Investigations) | 2 | 0
Gamma-glutamyltransferase increased (Investigations) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 7
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 9 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 5 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 3
Groin pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 0
Headache (Nervous system disorders) | 17 | 8
Dizziness (Nervous system disorders) | 9 | 5
Dysgeusia (Nervous system disorders) | 4 | 5
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 2
Cranial nerve disorder (Nervous system disorders) | 2 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 2
Paraesthesia (Nervous system disorders) | 2 | 0
Peripheral motor neuropathy (Nervous system disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 12 | 8
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5 | 4
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 1
Exfoliative rash (Skin and subcutaneous tissue disorders) | 3 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 3 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 12
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 8 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 6 | 7
Sinusitis (Infections and infestations) | 2 | 7
Urinary tract infection (Infections and infestations) | 2 | 2
Rhinitis (Infections and infestations) | 3 | 0
Viral infection (Infections and infestations) | 2 | 1
Ear infection (Infections and infestations) | 2 | 0
Influenza (Infections and infestations) | 2 | 0
Proteinuria (Renal and urinary disorders) | 5 | 8
Pollakiuria (Renal and urinary disorders) | 4 | 0
Haematuria (Renal and urinary disorders) | 2 | 1
Nocturia (Renal and urinary disorders) | 3 | 0
Anxiety (Psychiatric disorders) | 2 | 5
Insomnia (Psychiatric disorders) | 4 | 3
Depression (Psychiatric disorders) | 2 | 3
Confusional state (Psychiatric disorders) | 3 | 1
Hypothyroidism (Endocrine disorders) | 4 | 9
Adrenal insufficiency (Endocrine disorders) | 0 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 5
Anaemia (Blood and lymphatic system disorders) | 2 | 1
Contusion (Injury, poisoning and procedural complications) | 3 | 3
Excoriation (Injury, poisoning and procedural complications) | 0 | 2
Thermal burn (Injury, poisoning and procedural complications) | 2 | 0
Periorbital oedema (Eye disorders) | 3 | 0
Eye pain (Eye disorders) | 2 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 3
Atrial fibrillation (Cardiac disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.